CLINICAL TRIAL: NCT01661881
Title: A Phase II Study of Rituximab/Bendamustine Followed by Rituximab/Cytarabine for Untreated Mantle Cell Lymphoma
Brief Title: Rituximab/Bendamustine + Rituximab/Cytarabine for Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Philippe Armand, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-168
Record Dates: First submitted 2012-07-15; First posted 2012-08-10 (Estimated); Results first posted 2017-01-12 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Mantle Cell Lymphoma
Keywords: Newly diagnosed
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Rituximab; Bendamustine Hydrochloride; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RB/RC (Experimental): Patients received 3 cycles of outpatient RB (rituximab 375 mg/m2 day 1, bendamustine 90 mg/m2 days 1 and 2 of a 4-week cycle), followed by interim CT restaging. Patients with progressive disease (PD) went off study. Those with stable disease (SD) or better went on to receive three cycles of inpatient RC (rituximab 375 mg/m2 day 1, cytarabine 3 g/m2 every 12 h for 4 doses). The cytarabine was dose reduced to:
  1. 2 g/m2 for age >60 years old, creatinine 114.9-176.8 lmol/l (for patients ≤60 years old), and pre-existing neurotoxicity;
  2. 1.5 g/m2 for age >60 years old AND creatinine 114.9-176.8 lmol/l, or for age >60 years old AND pre-existing neurotoxicity;
  3. 1 g/m2 for age > 60 years old AND creatinine 114.9-176.8 lmol/l AND pre-existing neurotoxicity.
  Stem cell mobilization and collection, ASCT and post-transplantation supportive care were performed per institutional standard and not as part of this study.
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Cytarabine

INTERVENTIONS:
Drug: Rituximab
  Other Names: Rituxan
Drug: Bendamustine
  Other Names: Treanda
Drug: Cytarabine
  Other Names: Depocyt

SUMMARY:
Mantle cell lymphoma (MCL) is not curable with conventional therapy. This study sought to improve upon standard of care in newly diagnosed, untreated MCL patients who were transplant-eligible using drugs already established as active in MCL. The combination of Rituximab-Bendamustine followed by Rituximab-Cytarabine (RB/RC) was expected to maximize pre-ASCT complete response (CR) rate compared to historical rates approximating 55% with tolerable toxicity.

DETAILED DESCRIPTION:
This was a PII single-arm design to determine whether the regimen looked promising for further study.

Primary Objective

• To evaluate the efficacy of an alternating regimen of Rituximab-Bendamustine and Rituximab-Cytarabine (RB/RC) using the CR/Cru rate.

Secondary Objectives

* To assess safety.
* To estimate the rate of complete remission (CR), unconfirmed CR (CRu), partial remission (PR), stable disease (SD) and progressive disease (PD).
* To estimate the rate of successful stem cell mobilization after RB/RC in responding patients.
* To estimate the proportion of patients who can successfully complete the regimen and proceed to autologous stem cell transplantation (ASCT).
* To estimate the rate of neutrophil and platelet engraftment after ASCT.
* To estimate the CR/CRu and PR rate for patients with blastoid variant MCL.
* To estimate the rate of minimal residual disease (MRD)-negativity at treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Mandatory pathologic review of the diagnostic specimen(s) at Brigham and Women's Hospital or Massachusetts General Hospital
* Measurable disease
* Candidate for ASCT

Exclusion Criteria:

* Prior anti-lymphoma therapy
* Pregnant or breastfeeding
* Hypersensitivity to rituximab
* Uncontrolled intercurrent illness
* Receiving other study agents
* HIV positive on combination antiretroviral therapy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08-16 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2030-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Armand, MD, PhD, Study Chair — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Armand P, Redd R, Bsat J, Mayuram S, Giardino A, Fisher DC, LaCasce AS, Jacobson C, Davids MS, Brown JR, Weng L, Wilkins J, Faham M, Freedman AS, Joyce R, Jacobsen ED. A phase 2 study of Rituximab-Bendamustine and Rituximab-Cytarabine for transplant-eligible patients with mantle cell lymphoma. Br J Haematol. 2016 Apr;173(1):89-95. doi: 10.1111/bjh.13929. Epub 2016 Jan 5. PMID 26729345
- [Result] Merryman RW, Edwin N, Redd R, Bsat J, Chase M, LaCasce A, Freedman A, Jacobson C, Fisher D, Ng S, Crombie J, Kim A, Odejide O, Davids MS, Brown JR, Jacene H, Cashen A, Bartlett NL, Mehta-Shah N, Ghobadi A, Kahl B, Joyce R, Armand P, Jacobsen E. Rituximab/bendamustine and rituximab/cytarabine induction therapy for transplant-eligible mantle cell lymphoma. Blood Adv. 2020 Mar 10;4(5):858-867. doi: 10.1182/bloodadvances.2019001355. PMID 32126141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from August 2012 through March 2014.
Groups:
- RB/RC: Patients received 3 cycles of outpatient RB (rituximab 375 mg/m2 day 1, bendamustine 90 mg/m2 days 1 and 2 of a 4-week cycle), followed by interim CT restaging. Patients with progressive disease (PD) went off study. Those with stable disease (SD) or better went on to receive three cycles of inpatient RC (rituximab 375 mg/m2 day 1, cytarabine 3 g/m2 every 12 h for 4 doses). The cytarabine was dose reduced to:
  1. 2 g/m2 for age >60 years old, creatinine 114.9-176.8 lmol/l (for patients ≤60 years old), and pre-existing neurotoxicity;
  2. 1.5 g/m2 for age >60 years old AND creatinine 114.9-176.8 lmol/l, or for age >60 years old AND pre-existing neurotoxicity;
  3. 1 g/m2 for age > 60 years old AND creatinine 114.9-176.8 lmol/l AND pre-existing neurotoxicity.
Period: Overall Study
Arm/Group | RB/RC
Started | 23
Completed | 22
Not Completed | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | RB/RC
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 57 [42 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23
MIPI at Diagnosis [Count of Participants; unit: Participants] — The MIPI (Mantle Cell Lymphoma international prognostic index) (Hoster et al, 2008) is a risk index based on clinical characteristics (eg, LDH, white blood count, etc). Patients with higher MIPI scores tend to have a worse prognosis with frontline therapy.
  Participants
    Low | 16
    Intermediate | 5
    High | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR) Rate After 6 Cycles
Description: The CR rate is defined as the proportion of patients who after 6 cycles of therapy achieve complete remission based on the International Working Group (IWG) Criteria (Cheson et al, 1999), using CT scans. CR or CRu (CR unconfirmed) by CT scans was defined by standard IWG criteria, ie resolution of all abnormal adenopathy and organomegaly, and clearance of marrow disease when present at baseline.
Time Frame: Disease was assessed after three- and six-cycles of therapy, up to approximately 25 weeks. All patients completed 6 cycles of therapy with a cycle duration of 28 days.
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | RB/RC
Number analyzed (Participants) | 23
proportion of participants | .96 [.81 to 1.0]

2. Secondary Outcome: 1 Year Progression-Free Survival
Description: 1-year progression-free survival is the probability of patients remaining alive and progression-free at 1 year from study entry estimated using Kaplan-Meier methods. Disease progression was based on the International Working Group (IWG) Criteria (Cheson et al, 1999).
Time Frame: Disease was assessed after three- and six-cycles of therapy and in long-term follow-up per standard practice every 6 months until the earliest of relapse, death or 5 years. Median follow-up in this study cohort was 13 months.
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number (90% Confidence Interval); unit: probability
Arm/Group | RB/RC
Number analyzed (Participants) | 23
probability | .96 [.73 to .99]

3. Secondary Outcome: Autologous Stem Cell Transplant (ASCT) Rate
Description: ASCT rate is the proportion of patients who completed therapy and proceeded to autologous stem cell transplant (ASCT)
Time Frame: All patients were followed for continuation to ASCT upon completion of induction therapy. Patients usually proceed to ASCT within 3 months of completing induction.
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | RB/RC
Number analyzed (Participants) | 23
proportion of participants | .91 [.75 to .98]

ADVERSE EVENTS:
Time Frame: Assessed throughout the treatment period, from time of first dose and up to day 30 post-treatment, ie approximately 26 weeks. All patients received 6 cycles of therapy with protocol cycle duration of 28 days.
Description: Maximum grade toxicity by type was first calculated including only events with treatment-attribution of possible, probable or definite. Serious AEs and Other AEs were defined as treatment-related grade 3-5 events and grade 1-2 events, respectively, per CTCAEv4. No further data is available to specify classification of other beyond the general term.
Arm/Group | RB/RC
Serious Adverse Events (participants affected / at risk) | 15/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RB/RC (N=23)
Anemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 2
Sepsis (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 11
Neutrophil count decreased (Investigations) | 8
Platelet count decreased (Investigations) | 2
White blood cell decreased (Investigations) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RB/RC (N=23)
Anemia (Blood and lymphatic system disorders) | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Eye disorders - Other (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 19
Fever (General disorders) | 2
Infusion related reaction (General disorders) | 2
Irritability (General disorders) | 1
Pain (General disorders) | 2
General disorders and administration site conditions - Other (General disorders) | 1
Immune system disorders - Other (Immune system disorders) | 1
Mucosal infection (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 2
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 10
White blood cell decreased (Investigations) | 3
Investigations - Other (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4
Hypotension (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No